CLINICAL TRIAL: NCT05663879
Title: Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Characteristics of ID120040002 in Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetic and Pharmacodynamic of ID120040002 in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ID120040002-GERD-101
Record Dates: First submitted 2022-11-23; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- ID120040002 A mg (Experimental): Single dose 8 volunteers will be administered ID120040002 Amg or placebo comparators (ID120040002: placebo = 6:2)
  Interventions: Drug: ID120040002; Drug: Placebo comparator
- ID120040002 Bmg (Experimental): Single dose 8 volunteers will be administered ID120040002 Bmg or placebo comparators (ID120040002: placebo = 6:2)
  Interventions: Drug: ID120040002; Drug: Placebo comparator
- ID120040002 Cmg (Experimental): Single dose 8 volunteers will be administered ID120040002 Cmg or placebo comparators (ID120040002: placebo = 6:2)
  Interventions: Drug: ID120040002; Drug: Placebo comparator
- ID120040002 Dmg (Experimental): Period1:
  Single dose 8 volunteers will be administered ID120040002 Dmg or placebo comparators (ID120040002: placebo = 6:2)
  Period2:
  Single dose 8 volunteers will be administered ID120040002 Dmg or placebo comparators (ID120040002: placebo = 6:2)
  Interventions: Drug: ID120040002; Drug: Placebo comparator
- ID120040002 Emg (Experimental): Single dose 8 volunteers will be administered ID120040002 Emg or placebo comparators (ID120040002: placebo = 6:2)
  Interventions: Drug: ID120040002; Drug: Placebo comparator
- ID120040002 Fmg (Experimental): Multiple dose 10 volunteers will be administered ID120040004 F mg or placebo comparators (ID120040002: placebo: 8:2)
  Interventions: Drug: ID120040002; Drug: Placebo comparator
- ID120040002 Gmg (Experimental): Multiple dose 10 volunteers will be administered ID120040004 G mg or placebo comparators (ID120040002: placebo: 8:2)
  Interventions: Drug: ID120040002; Drug: Placebo comparator
- ID120040002 Hmg (Experimental): Multiple dose 10 volunteers will be administered ID120040004 H mg or placebo comparators (ID120040002: placebo: 8:2)
  Interventions: Drug: ID120040002; Drug: Placebo comparator
- ID120040002 Img (Experimental): Multiple dose 10 volunteers will be administered ID120040004 I mg or placebo comparators (ID120040002: placebo: 8:2)
  Interventions: Drug: ID120040002; Drug: Placebo comparator
- Compound-X Jmg (Active Comparator): Multiple dose 8 volunteers will be administered compound-X J mg
  Interventions: Drug: Compound-X

INTERVENTIONS:
Drug: ID120040002 — Drug: ID120040002
  Arms: ID120040002 A mg; ID120040002 Bmg; ID120040002 Cmg; ID120040002 Dmg; ID120040002 Emg; ID120040002 Fmg; ID120040002 Gmg; ID120040002 Hmg; ID120040002 Img
Drug: Compound-X — Drug: Compound-X
  Arms: Compound-X Jmg
Drug: Placebo comparator — Placebo comparator
  Arms: ID120040002 A mg; ID120040002 Bmg; ID120040002 Cmg; ID120040002 Dmg; ID120040002 Emg; ID120040002 Fmg; ID120040002 Gmg; ID120040002 Hmg; ID120040002 Img

SUMMARY:
A Randomized, Double-blinded, Partial-open, Placebo and Active-controlled, Single and Multiple Dose-escalation Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Characteristics of ID120040002 in Healthy Volunteers

DETAILED DESCRIPTION:
To evaluate the safety, tolerability, and pharmacokinetic characteristics and to explore pharmacodynamic characteristics and food effects after single and multiple doses of ID120040002 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have a body weight of ≥50.0 kg to ≤90.0 kg, and Body Mass Index (BMI) of ≥18.0 kg/m2 to ≤27.0 kg/m2
* Subjects who have decided to voluntarily participate and consented in writing to comply with the precautions after listening to a detailed explanation of this clinical study
* Subjects who consent to use contraceptive methods* accepted in this trial with their partners and not to donate sperm until 90 days and eggs until 28 days after the administration of the last dose of the IP from the time of written consent.

Exclusion Criteria:

* Subjects with a history of clinically significant cardiovascular, respiratory, renal, endocrine, hematological, gastrointestinal, central nervous system, urinary, musculoskeletal and psychological disorders or malignant tumor, or current active diseases (however, subjects may be enrolled if the disease is completely recovered and does not affect the current health status)
* Subjects with a history of gastrointestinal disease (Crohn's disease, ulcer, acute or chronic pancreatitis, hypochlorhydria, achlorhydria, etc.) or gastrointestinal surgery (excluding simple appendectomy and herniotomy) that can affect the absorption of the investigational product
* Subjects who have received the therapy for peptic ulcer, esophageal disease or Zollinger-Ellison syndrome within 90 days prior to the administration of the IP, or have clinically suspected symptoms of such diseases
* Subjects who have received H. pylori eradication therapy within 6 months, or have positive result for H. pylori test at screening

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Serious Adverse Events (SAEs) | From Screening (Day -28 to -3) until termination (approximately Day 8 for SAD and Day 14 for MAD)
  To evaluate the safety and tolerability of single and multiple ascending doses of ID120040002 in healthy participants.
Number of participants with Adverse Events (AEs) | From Screening (Day -28 to -3) until termination (approximately Day 8 for SAD and Day 14 for MAD)
  To evaluate the safety and tolerability of single and multiple ascending doses of ID120040002 in healthy participants.
Percentage of subjects with clinically significant change from baseline in vital signs | From Screening (Day -28 to -3) until termination (approximately Day 8 for SAD and Day 14 for MAD)
Percentage of subjects with clinically significant change from baseline in electrocardiogram (ECG) | From Screening (Day -28 to -3) until termination (approximately Day 8 for SAD and Day 14 for MAD)

CONTACTS AND LOCATIONS:
Overall Officials: SeungHwan Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea